CLINICAL TRIAL: NCT03246867
Title: The Acute Effects of Different Stretching Methods on Posterior Shoulder Tightness, Pain, Joint Range of Motion, Subacromial Space and Strength in Individuals Having Subacromial Impingement Syndrome With Glenohumeral Internal Rotation Deficit
Brief Title: The Acute Effects of Different Stretching Methods in Individuals With Subacromial Impingement Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Halime Ezgi TÜRKSAN, Research Assistant, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3418-GOA
Record Dates: First submitted 2017-08-08; First posted 2017-08-11 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Subacromial Impingement Syndrome; Glenohumeral Internal Rotation Deficit
Keywords: isolytic stretching; static stretching; Glenohumeral Internal Rotation Deficit
MeSH Terms: conditions — Shoulder Impingement Syndrome | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: There are 3 groups. First group will receive isolytic stretching in modified cross body position. Second group will receive static stretching in modified cross body position. The stretching exercise will be applied five times each for 15 seconds. After each stretching there will be a resting period for 5 seconds. Control group will receive no stretching. They will be handed a brochure about the stretching techniques and its role in injury prevention. Isolytic and static stretching groups will be evaluated before and just after stretching exercise. Control group will be evaluated for the first time and then will be passively waited until the duration of the stretching exercise program (approximately 4-5 min). Afterwards, second evaluation will be performed.
Who Masked: Participant
Masking Description: All of participants must have subacromial impingement syndrome with glenohumeral internal rotation deficit.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Isolytic stretching group (Experimental): The participants in this group will receive isolytic stretching in modified cross body position.
  Interventions: Other: Isolytic stretching group
- Static stretching group (Experimental): The participants in this group will receive static stretching in modified cross body position.
  Interventions: Other: Static stretching group
- Control group (Active Comparator): The participants in this group will receive no stretching. They will only be evaluated.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Isolytic stretching group — In modified cross body position, isolytic stretching exercises will perform five times each for 15 seconds. After each stretching patient will rest for 5 seconds. When the patient contracts the agonist muscle group with 20% muscle force, the agonist muscle group is stretched at the same time for 2-4 seconds. Afterwards active-assistive stretching is done. Evaluations will be done before and just after stretching exercise.
  Arms: Isolytic stretching group
Other: Static stretching group — In modified cross body position, active-assistive static stretching exercises will be performed 5 times each for 15 seconds. This stretching exercise is performed 5 times with 5 seconds intervals. Evaluations will be done before and just after stretching exercise.
  Arms: Static stretching group
Other: Control group — Control group will receive no stretching. They will be handed a brochure about the stretching techniques and its role in injury prevention. Control group will be evaluated for the first time and then will be passively waited until the duration of the stretching exercise program (approximately 4-5 min). Afterwards, second evaluation will be performed.
  Arms: Control group

SUMMARY:
The purpose of this study is to investigate and compare the acute effects of isolytic and static stretching training in individuals having subacromial impingement syndrome with glenohumeral internal rotation deficit. Isolytic group will receive isolytic stretching in modified cross body position. Static group will receive static stretching in modified cross body position. Stretching groups will be evaluated before and just after stretching exercise. Control group will receive no stretching. Control group will be evaluated for the first time and then will be waited until the duration of the stretching exercise program. Afterwards, second evaluation will be performed

DETAILED DESCRIPTION:
There is no information in literature about the acute effects of isolytic stretching exercise in individuals having subacromial impingement syndrome with glenohumeral internal rotation deficit. The purpose of this study is to investigate and compare the acute effects of isolytic and static stretching training in individuals having subacromial impingement syndrome with glenohumeral internal rotation deficit.

In modified cross body position, static stretching group will perform active-assistive static stretching by the physiotherapist whereas isolytic stretching group will perform active-assistive isolytic stretching. Stretching exercises will be applied five times each for 15 seconds. After each stretching there will be a resting period for 5 seconds. Control group will receive no stretching. They will be handed a brochure about the stretching techniques and its role in injury prevention. Isolytic and static stretching groups will be evaluated before and just after stretching exercise. Control group will be evaluated for the first time and then will be passively waited until the duration of the stretching exercise program (approximately 4-5 min). Afterwards, second evaluation will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of subacromial impingement syndrome
* Glenohumeral internal rotation range of motion of the affected shoulder should be less than other shoulder and bilateral shoulder internal rotation range of motion difference should be ≥15 º
* Pain with resisted arm elevation or external rotation as well as a minimum of 3 of 5 positive subacromial impingement syndrome tests, painful arc, pain or weakness with resisted external rotation, Neer, Hawkins and Jobe tests .
* Ability to complete the entire study procedure

Exclusion Criteria:

* An inability to elevate the involved arm greater than 140 degree in the scapular plane
* A 50% limitation of passive shoulder range of motion in >2 planes of motion
* Pain >7/10
* A history of fracture to the shoulder girdle
* Systemic musculoskeletal disease
* History of shoulder surgery,
* Glenohumeral instability (positive apprehension, relocation or positive sulcus test) or positive findings for a full thickness rotator cuff tear (positive lag sign, positive drop arm test or marked weakness with shoulder external rotation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2020-01-02 (Actual)

PRIMARY OUTCOMES:
Shoulder internal rotation range of motion | Baseline and just after stretching exercise
  Change of shoulder internal rotation range of motion (with bubble inclinometer)

SECONDARY OUTCOMES:
Posterior shoulder tightness | Baseline and just after stretching exercise
  Change of posterior shoulder tightness (with bubble inclinometer)
Concentric strength | Baseline and just after stretching exercise
  Change of trapezius muscles, rotattor cuff muscles concentric strength (in kg, with hand held dynamometer)
Eccentric strength | Baseline and just after stretching exercise
  Change of shoulder abduction and external rotation eccentric strength (in kg, with hand held dynamometer)
Subacromial space | Baseline and just after stretching exercise
  Change of subacromial space ( with Ultrasound)
Pain | Baseline and just after stretching exercise
  Change of visual analog scale score in activity and rest
Shoulder external rotation range of motion | Baseline and just after stretching exercise
  Change of shoulder external rotation range of motion (with bubble inclinometer)

CONTACTS AND LOCATIONS:
Overall Officials: Sevgi Sevi YESILYAPRAK, PhD, Study Director — Dokuz Eylul University; Damla GULPINAR, MS, Study Director — Izmir Katip Celebi University; Mehmet ERDURAN, MD, Study Director — Dokuz Eylul University; Cem OZCAN, MD, Study Director — Izmır Katip Celebi University Atatürk Training and Research Hospital
Locations (1):
- Dokuz Eylül University, Izmir, Turkey (Türkiye)